CLINICAL TRIAL: NCT00469261
Title: Tetracycline (Doxycycline) In Patients With Large Acute Myocardial Infarction TO Prevent Left Ventricular Remodeling. TIPTOP Study
Brief Title: Tetracycline (Doxycycline) and Post Myocardial Infarction Remodeling
Acronym: TIPTOP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Careggi Hospital (Other)
Responsible Party: Principal Investigator, David Antoniucci, MD, Careggi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIP-TOP
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Myocardial Infarction; Left Ventricular Remodeling
Keywords: Myocardial infarction; Ventricular remodeling; Matrix metalloproteinases; Doxycycline
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Experimental): Active drug 100 mg bid for seven days in pts with AMI treated with Primary PCI and current medical therapy
  Interventions: Drug: Doxycycline
- Standard Therapy (Active Comparator): Pts with AMI treated with Primary PCI and current medical therapy
  Interventions: Drug: Current medical therapy for AMI

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg bid for seven days after enrollment
  Arms: Doxycycline
Drug: Current medical therapy for AMI — Current medical therapy for AMI
  Arms: Standard Therapy

SUMMARY:
The aim of the study is to assess the efficacy of an antibiotic treatment with tetracycline (doxycycline) in the early stage of large reperfused acute myocardial infarction (AMI), in preventing left ventricular (LV) remodeling.

DETAILED DESCRIPTION:
A myocardial interstitial matrix, that provides structural support and integrity to the myocardium, is a key element to determine post infarction left ventricular remodeling (LVR).

The metalloproteinases (MMPs), an enzymatic system secreted in the extracellular medium by macrophages, has been shown to be able to degrade the most important extracellular matrix components.

Various animal experimental models have demonstrated that MMP specific inhibition in the first phase of myocardial infarction is able to contrast LVR. Doxycycline, a member of the tetracyclines, has been shown to block various inflammation mediators and to attenuate MMP-2 and MMP-9 expression and activity at a sub-antimicrobial dosage. Some experimental studies on rat models have suggested an anti-remodeling effect of doxycycline in myocardial infarction.

In the present study we want to evaluate if a treatment with doxycycline (100 mg b.i.d.) in the first seven days after a reperfused large (ejection fraction less than 40%) acute myocardial infarction, is effective in preventing six-month LVR.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Left ventricular ejection fraction less than 40%

Exclusion Criteria:

* No written consensus
* Allergy to tetracycline
* Mechanical complication of AMI
* Previous myocardial infarction
* Valvular and/or myocardiopathy known or suspected
* Renal failure (creatinine above 2 mg/dL)
* Connective tissue disease
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Reduction of LV dilation (six months versus baseline LV end-diastolic volume index by 2D-echocardiogram [echo]) more than 50% in the treated group in comparison to the placebo group | 6 months

SECONDARY OUTCOMES:
Evaluation of the time course of MMPs and their inhibitors in relation to left ventricular remodeling | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Cerisano, MD, Principal Investigator — Careggi Hospital, Florence, Italy; David Antoniucci, MD, Study Director — Careggi Hospital, Florence, Italy; Piergiovanni Buonamici, MD, Study Chair — Careggi Hospital, Florence, Italy; Emilio V Dovellini, MD, Study Chair — Careggi Hospital, Florence, Italy; Alberto Santini, MD, Study Chair — Careggi Hospital, Florence, Italy; Umberto Signorini, MD, Study Chair — Careggi Hospital, Florence, Italy; Nazario Carrabba, MD, Study Chair — Careggi Hospital, Florence, Italy; Paolo D Pucci, MD, Study Chair — Careggi Hospital, Florence, Italy; Renato Valenti, MD, Study Chair — Careggi Hospital , Florence, Italy

REFERENCES:
- [Derived] Cerisano G, Buonamici P, Valenti R, Sciagra R, Raspanti S, Santini A, Carrabba N, Dovellini EV, Romito R, Pupi A, Colonna P, Antoniucci D. Early short-term doxycycline therapy in patients with acute myocardial infarction and left ventricular dysfunction to prevent the ominous progression to adverse remodelling: the TIPTOP trial. Eur Heart J. 2014 Jan;35(3):184-91. doi: 10.1093/eurheartj/eht420. Epub 2013 Oct 8. PMID 24104875